CLINICAL TRIAL: NCT04299334
Title: A Novel Adjustable Neochordae Technique in Mitral Valve Repair
Brief Title: Neochordae Technique in Mitral Valve Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Yosry Mahmoud Thakeb, Principal Investigator, National Heart Institute, Egypt
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHI-MR-001
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Mitral Valve Prolapse; Mitral Regurgitation
Keywords: neochordae; Mitral valve repair
MeSH Terms: conditions — Mitral Valve Prolapse; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: adjustable neochordae Technique — Classic ring annuloplasty will be done using Carpentier or physio ring, then neochordal placement will be done using the looping technique. The length of the chordae is adjusted to achieve the optimal length.
  In this study, Surgeons use relatively short loops because of the augmentation of the length with extra loops suspended with Gortex. Placement of at least 8-12 chordae of the corresponding heads of the papillary muscle tip to achieve proper management of the prolapse and longevity of the repair.

SUMMARY:
Mitral valve (MV) repair has turned into a preferable option for surgeons over the MV replacement. Since the 1960s, Surgeons use this technique for more efficiency and durability. On the other hand, the proper determination of length and placement of artificial neochordae is still a challenge beyond this technique. These challenges are still a vital area for research and debate between surgeons and researchers.

In our novel technique,Investigators are not depending either on the preoperative investigations or intraoperative reference chordae in the adjustment of the optimal length of the neochordae, however, Researchers depend on the personal adjustment of the chordal length to the prolapsed scallop.

DETAILED DESCRIPTION:
Mitral regurgitation (prolapse) and mitral stenosis are examples of diseases that affect the mitral valve. In mitral regurgitation, the leaflets do not close tightly and sway up and down allowing the blood to flow backward from the left ventricle into the left atrium. on the other hand, the mitral stenosis is caused by folding of thick leaflets of the valve which fuses together leading to low blood flow from the left atrium into the left ventricle and these cases are excluded from our trial. In mitral regurgitation, Surgeons prefer the mitral valve repair over the mitral valve replacement, But still, there are a lot of challenges towards this technique.

For decades, Surgeons used a lot of techniques to determine the length of neochordae includes that:

Determination of neochordal length by transoesophageal echocardiography or by using a landmark as a direct measurement. Previously, the surgeon applying the fixed loop length technique by using a custom-made caliper, and on the distance between the edge of a non-prolapsing segment and the tip of the papillary muscle (usually P1) to define the correct loop length. There are different types of papillary muscle and chordae as regards the shape, morphology, and length. So this reference distance is not fixed.

Adjusting neochordal length according to valve function. Length is chosen when the regurgitation is completely removed. Existing of a large number of neochordae will make this process more complex for the surgeon to decide.

Mitral valve (MV) repair has turned into a preferable option for surgeons over the MV replacement. Since the 1960s, Surgeons use this technique for more efficiency and durability. On the other hand, the proper determination of length and placement of artificial neochordae is still a challenge beyond this technique. These challenges are still a vital area for research and debate between surgeons and researchers.

In our novel technique, Investigators are not depending either on the preoperative investigations or intraoperative reference chordae in the adjustment of the optimal length of the neochordae, however, Researchers depend on the personal adjustment of the chordal length to the prolapsed scallop.

ELIGIBILITY:
Inclusion Criteria:

* Prolapsed or ruptured chordae
* Either degenerative or ischemic

Exclusion Criteria:

* Patient with redo Mitral Valve surgery
* Patient with severe rheumatic mitral stenosis (MS).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
competency of mitral valve repair | 6 months follow up
  by using the transthoracic echocardiography or the trans-esophageal echo to measure the mitral valve competency and the degree of mitral regurge.

CONTACTS AND LOCATIONS:
Overall Officials: Yosry Thakeb, M.D., Principal Investigator — Cardiothoracic Surgery Department, National Heart Institute, Giza, Egypt.; Amr Zaher, M.D., Principal Investigator — Adjunct Professor, Biomedical sciences program, Zewail City of Science and Technology
Locations (1):
- Yosry Mahmoud Thakeb, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided